CLINICAL TRIAL: NCT05591560
Title: The Possible Effect of Itraconazole as add-on Therapy to Paclitaxel and Carboplatin on the Treatment Outcome in Patients With Advanced Ovarian Cancer
Brief Title: Itraconazole in Advanced Ovarian Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ahmed Ezzat Saad Besheir, Clinical Pharmacist, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35929/10/22
Record Dates: First submitted 2022-10-17; First posted 2022-10-24 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Ovarian Carcinoma
Keywords: Itraconazole; Paclitaxel; Carboplatin; Chemotherapy; Epithelial; Ovarian; Carcinoma
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma | interventions — Itraconazole

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I Placebo group (Placebo Comparator): Group I (Placebo group; n=33) which will be treated with chemotherapy which includes paclitaxel 60 mg/m2 IV over 1 hour followed by carboplatin area under the curve 2 (AUC 2) IV over 30 minutes Day 1, 8, and 15 which will be repeated every 21 days for 6 cycles 12 plus 4 placebo capsules for 5 days (two days before chemotherapy, the day of chemotherapy after receiving it, and two days after chemotherapy).
  Interventions: Drug: Placebo
- Group II Itraconazole group (Active Comparator): Group II: (Itraconazole group; n=33) which will be treated with chemotherapy which includes paclitaxel 60 mg/m2 IV over 1 hour followed by carboplatin AUC 2 IV over 30 minutes Day 1, 8, and 15 repeated every 21 days for 6 cycles 12 plus oral itraconazole 400 mg (4 capsules, each of 100 mg) for 5 days (two days before chemotherapy, the day of chemotherapy after receiving it, and two days after chemotherapy).
  Interventions: Drug: Itraconazole capsule

INTERVENTIONS:
Drug: Itraconazole capsule — Oral itraconazole 400 mg (4 capsules, each of 100 mg) for 5 days (two days before chemotherapy, the day of chemotherapy after receiving it, and two days after chemotherapy) Day 1, 8, and 15 repeated every 21 days for 6 cycles for group II
  Arms: Group II Itraconazole group
Drug: Placebo — 4 placebo capsules for 5 days (two days before chemotherapy, the day of chemotherapy after receiving it, and two days after chemotherapy) Day 1, 8, and 15 repeated every 21 days for 6 cycles for group I
  Arms: Group I Placebo group

SUMMARY:
This is a randomized, placebo controlled; parallel study that will be conducted on 66 female patients with advanced epithelial ovarian carcinoma (stage III and stage IV) to compare effect of adding Itraconazole to paclitaxel and carboplatin versus placebo to paclitaxel and carboplatin as regard overall response rate (ORR) and Disease control rate (DCR) and Quality of life (QOL) and the change in the serum concentrations of the biological markers.

DETAILED DESCRIPTION:
This is a randomized, placebo controlled; parallel study that will be conducted on 66 female patients with advanced epithelial ovarian carcinoma (stage III and stage IV). The staging of the disease will be done according to 8th edition of American Joint Committee on Cancer (AJCC), TNM staging. The patients will be recruited from Oncology Department, Tanta University Hospital. The patients will receive a combination of paclitaxel and carboplatin chemotherapy with or without itraconazole. Randomization will be carried out based on hospital admission days where the patients will be randomized into the following two groups to compare effect of adding Itraconazole to paclitaxel and carboplatin versus placebo to paclitaxel and carboplatin.

ELIGIBILITY:
Inclusion Criteria:

* Female patients Age >18 years old < 65 years old.
* Patients with histopathological and radiological based diagnosis of III, IV epithelial ovarian carcinoma according to 8th edition AJCC, primary tumor, regional nodes, metastasis (TNM) staging system.11
* Patients with Eastern Cooperative Oncology Group Performance Status of 0 or 1. 13
* Patients able to swallow and retain oral medications (without crushing, dissolving, or chewing tablets).
* Patients with adequate hematologic and organ function within 14 days before the first Cycle which can be defined by the following:

  * Neutrophils (absolute neutrophil count (ANC) >1.5 X 10^9/L).
  * Hemoglobin >9 g/dl.
  * Platelet count >100,000/L.
  * Serum albumin >3 g/dl.
  * Total bilirubin 1.5 ≤ of the upper limit of normal (ULN) and aspartate aminotransferase (AST) and alanine transaminase ( ALT) ≤ 2 of the upper limit of normal (ULN).
  * Serum creatinine ≤ 1.5 of the upper limit of normal (ULN) or estimated creatinine clearance >50 mL/min based on Cockcroft-Gault glomerular filtration rate estimation.

Exclusion Criteria:

* Presence of 2nd primary malignancy
* History of allergic reactions attributed to paclitaxel, carboplatin, and itraconazole or to compounds of similar chemical or biologic composition to itraconazole.
* Concurrent use of medications significantly affecting metabolism of itraconazole (certain anti-convulsants).
* Patients with hyperthyroidism (which would increase metabolism of itraconazole).
* Patients with grade ≥ 2 neuropathy.
* Patients with Uncontrolled, concurrent medical illness.
* Patients with active hepatitis or symptomatic liver disease.
* History of or current evidence of uncontrolled cardiac ventricular dysfunction (congestive heart failure) or patients with class III and class IV heart failure according to New York Heart Association (NYHA).
* Pregnant or lactating female .

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Measuring tumor response in epithelial ovarian carcinoma
Enrollment: 66 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The change between 2 groups in overall response rate and disease control rate | 1 week after the end of chemotherapy cycle 3 and 6 (each cycle is 21 days) and every 2 to 4 months after the end of 6 chemotherapy cycles (each cycle is 21 days) for 1 year
  The change between 2 groups in overall response rate and disease control rate using the Response Evaluation Criteria in Solid Tumors (RECIST), version. 1.1.

SECONDARY OUTCOMES:
The change in the serum concentrations of the biological markers (CA-125, VEGFR-2, P-glycoprotein). | 1 week after the end of chemotherapy cycle 3 and 6 (each cycle is 21 days) and every 2 to 4 months after the end of 6 chemotherapy cycles (each cycle is 21 days) for 1 year
  * Serum cancer antigen-125 (CA-125) level which will be assessed at baseline for all patients, after the third chemotherapy cycle and after the sixth chemotherapy cycle if it is positive at initial presentation.
  * Serum vascular endothelial growth factor receptor-2 (VEGFR-2) level by ELISA which will be assessed at baseline and after the sixth chemotherapy cycle.
  * Serum P-glycoprotein level by ELISA which will be assessed at baseline and after the sixth chemotherapy cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Tarek M Mostafa, Professor, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Faculty of Pharmacy, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goenka L, Dubashi B, Selvarajan S, Ganesan P. Use of "Repurposed" Drugs in the Treatment of Epithelial Ovarian Cancer: A Systematic Review. Am J Clin Oncol. 2022 Apr 1;45(4):168-174. doi: 10.1097/COC.0000000000000900. PMID 35320817
- [Background] Nunes M, Henriques Abreu M, Bartosch C, Ricardo S. Recycling the Purpose of Old Drugs to Treat Ovarian Cancer. Int J Mol Sci. 2020 Oct 20;21(20):7768. doi: 10.3390/ijms21207768. PMID 33092251
- [Background] Mohamed AW, Elbassiouny M, Elkhodary DA, Shawki MA, Saad AS. The effect of itraconazole on the clinical outcomes of patients with advanced non-small cell lung cancer receiving platinum-based chemotherapy: a randomized controlled study. Med Oncol. 2021 Feb 9;38(3):23. doi: 10.1007/s12032-021-01475-0. PMID 33559053
- [Background] Li CL, Fang ZX, Wu Z, Hou YY, Wu HT, Liu J. Repurposed itraconazole for use in the treatment of malignancies as a promising therapeutic strategy. Biomed Pharmacother. 2022 Oct;154:113616. doi: 10.1016/j.biopha.2022.113616. Epub 2022 Aug 30. PMID 36055112